CLINICAL TRIAL: NCT06164886
Title: Information Flow of Waiting List for Scheduled Surgical Admissions
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: LIDIA
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Chirurgical Intervention
MeSH Terms: interventions — Waiting Lists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sperimental: Patient on the waiting list for scheduled surgical admissions
  Interventions: Other: Waiting list

INTERVENTIONS:
Other: Waiting list — patient on the waiting list for scheduled surgical admissions

SUMMARY:
Definition and experimentation of the aforementioned information flow within the Regions participating in the three-year project, a Technical Subgroup was identified on a voluntary basis in charge of defining the design and following the experimental operational phases

ELIGIBILITY:
Inclusion Criteria:

* all adult patients

Exclusion Criteria:

* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients placed on the waiting list with the NHS for surgery scheduled at the centre
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Verification of the completeness of the data entered within the flow to guarantee ex Ante monitoring of the waiting list for scheduled surgical hospitalization | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes